CLINICAL TRIAL: NCT05680610
Title: Follow up of Moderate Aortic Regurge After Rhumatic Mitral Valve Replacement
Brief Title: Follow up of Moderate Aortic Regurge After Mitral Valve Replacement
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed wahba, Principle investigator, Assiut University
Other Study IDs: Assuit unimed
Record Dates: First submitted 2022-12-31; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Follow up of Moderate Aortic Regurge After Rheumatic Mitral Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim of the study is to follow of of moderate aortic regurge after mitral valve replacement to figure out if the aortic regurge has been improved or it is getting worse

DETAILED DESCRIPTION:
A considerable proportion of patients who require mitral valve replacement present with a coexisting pathology of the aortic valve (AV). Rheumatic fever remains the leading cause for combined disease (1) Early series found that one-third of rheumatic hearts exhibited involvement of both mitral and aortic valve. The rate increased to 99% when the follow-up period was extended to 20 years The treatment of choice in cases in which one of the valves is moderately affected is questionable. Because combined aortic and mitral valve replacement is usually associated with higher risk and poorer long-term survival than replacement of either of the two valves alone (2) In patients with moderate aortic regurgitation who undergo mitral valve surgery). according to 2021 ESC/EACTS Guidelines, the decision to treat the aortic valve is controversial, as data show that progression of moderate aortic regurgitation is very slow in patients without aortic dilation (3) in contrast , In 2020 AHA guidelines recommended concomitant aortic valve replacement for moderate aortic regurgitation in patients undergoing surgery for ascending aorta, coronary artery bypass grafting (CABG),or mitral valve surgery (4-10) Because of this is a point of conflict we aim in this study to evaluate the saftey to leave moderate aortic regurge without intertvention as regarding operative time ,postoperative morbidity and mortality and progression of aortic valve regurge.

ELIGIBILITY:
Inclusion Criteria:

* patients underwent mitral valve replacement for rheumatic heart disease and having moderate aortic valve regurge GRADE 2 in assuit university hospitals

Exclusion Criteria:

* non rhumatic heart disease ,severe aortic regurge ,moderately severe aortic regurge ,combined ischmic and valvular heart diseaese

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients who underwent mitral valve replacement with untrated concomitant moderate aortic regurge in Asyut university hospitals
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Comparison between pre operative degree of aortic regurge and Postoperative degree of aortic regurge after rheumatic mitral valve replacement | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: No